CLINICAL TRIAL: NCT03826485
Title: A Randomized, Open-label, Single-dose, Crossover Study to Compare Pharmacokinetics of PRIC and Pranlukast Dry Syrup in Healthy Male Volunteers
Brief Title: Safety, Pharmacokinetic Study of PRIC in Healthy Adult Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SamA Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRIC
Record Dates: First submitted 2016-12-28; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: Pranlukast hydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): Period 1: PRIC Period 2: Pranlukast hydrate
  Interventions: Drug: PRIC; Drug: Pranlukast hydrate
- B group (Experimental): Period 1: Pranlukast hydrate Period 2: PRIC
  Interventions: Drug: PRIC; Drug: Pranlukast hydrate

INTERVENTIONS:
Drug: PRIC — Pranlukast hydrate 50mg
  Other Names: PRIC 50mg
Drug: Pranlukast hydrate — Pranlukast hydrate 225mg/2.25g

SUMMARY:
The purpose of this study is Safety, Pharmacokinetic Study of PRIC

DETAILED DESCRIPTION:
1. To Compare Pharmacokinetics of PRIC and Pranlukast Dry Syrup
2. To evaluate the safety and tolerability of PRIC and Pranlukast Dry Syrup

ELIGIBILITY:
Inclusion Criteria:

* 19 to 45 years old healthy male subject at the screening
* Subject who is able to provide written informed consent and decided on his own participation after understanding fully to hear a detailed explanation in the clinical study

Exclusion Criteria:

* Subject with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption etc.
* Subjects with history of clinically significant allergy, cardiovascular, peripheral vascular, skin, mucocutaneous, ocular, ear, nose and throat (ENT), respiratory, musculoskeletal, infectious, gastrointestinal, liver, biliary, endocrine, renal, genitourinary, nervous, psychiatric, blood disorders, tumors, fractures or any other conditions

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-04-25 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) to last time point (t) | 0, 0.5, 0.75, 1, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10 and 12hours postdose
  Area under the PRIC/Pranlukast dry syrup concentration in blood-time curve from zero to the final
Maximum concentration of drug (Cmax) | 0, 0.5, 0.75, 1, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10 and 12hours postdose
  The maximum PRIC/Pranlukast dry syrup concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No